CLINICAL TRIAL: NCT02674009
Title: Non-Interventional Study to Investigate the Effectiveness, Safety and Utilization of Vismodegib on Locally Advanced Basal Cell Carcinoma Under Real World Conditions (NIELS)
Brief Title: Observational Study to Determine the Effectiveness and Safety of Vismodegib (Erivedge®) in Participants With Locally Advanced Basal Cell Carcinoma (laBCC)
Acronym: NIELS
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29670
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- laBCC Participants: Participants with laBCC who received at least one dose of Vismodegib in routine clinical practice for 32 months (between 02 Aug 2013 and 31 Mar 2016).
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — Participants with laBCC will receive a dosing of Vismodegib in accordance with local clinical practice and local labeling.
  Other Names: ERIVEDGE

SUMMARY:
The primary purpose for this multi-center, non-interventional study is to evaluate the duration of response defined as duration from first documented response of complete response (CR) or partial response (PR) until disease progression (as determined by the treating physician) for participants with laBCC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed IaBCC (inappropriate for surgery or radiotherapy)
* Participant is not included in any other trial
* Male or female participants are included in the pregnancy prevention program

Exclusion Criteria:

Participants for whom treatment with Vismodegib is contraindicated according to the SmPC, which has been in effect at the time of treatment with Vismodegib, including:

* Hypersensitivity to the active substance or to any of the excipients
* Women who are pregnant or breastfeeding
* Women of childbearing potential who do not comply with the Vismodegib Pregnancy Prevention Programme
* Coadministration of St John's wort (Hypericum perforatum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving/having received Vismodegib for treatment of laBCC according to the German label and in line with the current Summary of Product Characteristics (SmPC) and who have no contraindication to Vismodegib therapy as per the local label are eligible for this non-interventional study if written informed consent is provided.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Duration of Response, Defined as the Time from the First Assessment of CR or PR until Disease Progression or Death from any Cause, Whichever Occurs First | From first objective response until disease progression or death from any cause, up to 3 years

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response (CR or PR) as Determined by the Physician | From date of first therapy until disease progression or death, whichever occurs first (up to 3 years)
Percentage of Participants with Disease Control (CR, PR, or Stable Disease) | From date of first therapy until disease progression or death, whichever occurs first (up to 3 years)
Percentage of Participants with Disease Reccurence, Defined as Participants who Achieve CR and later Progress | From date of first therapy until disease progression or death, whichever occurs first (up to 3 years)
Progression-Free Survival, Evaluated According to Physician's Assessments | From the date of first therapy to disease progression or death from any cause, up to 3 years
Overall Survival | From the date of the first therapy to death from any cause, up to 3 years
Time to Response | From the date of first therapy to first confirmed CR or PR whichever occurs first, up to 3 years
Percentage of Participants with Adverse Events | From Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Klinik Johann Wolfgang von Goethe Uni; Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt, Germany